CLINICAL TRIAL: NCT03275701
Title: Phase IV, Single-Arm, Open-Label Study Evaluating Bone Mineral Density in HIV-1-Infected Adults ≥50 Years Old Switching From EVG/COBI/FTC/TAF (Genvoya) or EVG/COBI/FTC/TDF (Stribild) to ABC/DTG/3TC (Triumeq)
Brief Title: Evaluating BMD in Participants ≥50 Years Old Switching From EVG/COBI/FTC/TAF or EVG/COBI/FTC/TDF to ABC/DTG/3TC
Acronym: STRUCTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mills Clinical Research (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Anthony Mills MD, Clinical Research Director, Mills Clinical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205773
Record Dates: First submitted 2016-07-22; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triumeq (Other): Single Arm, Open Label
  Interventions: Drug: Triumeq

INTERVENTIONS:
Drug: Triumeq — Open Label, Switch to Triumeq (ABC/DTG/3TC)

SUMMARY:
Phase IV, Single-Arm, Open-Label Study Evaluating Bone Mineral Density in HIV-1-Infected Adults ≥50 Years Old Switching from EVG/COBI/FTC/TAF (Genvoya) or EVG/COBI/FTC/TDF (Stribild) to ABC/DTG/3TC (Triumeq)

DETAILED DESCRIPTION:
Phase IV, Single-Arm, Open-Label Study Evaluating Bone Mineral Density in HIV-1-Infected Adults ≥50 Years Old Switching from EVG/COBI/FTC/TAF (Genvoya) or EVG/COBI/FTC/TDF (Stribild) to ABC/DTG/3TC (Triumeq)

To evaluate the impact on BMD, as measured by DEXA over 48 weeks, of switching from an INSTI-based regimen with either TDF or TAF to a regimen of ABC/DTG/3TC (administered as commercial Triumeq) in chronic HIV-infected patients over the age of 50

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV-1 infection;
2. At least 50 years of age;
3. Currently on a stable antiretroviral regimen (for ≥3 months preceding Screening) of either EVG/COBI/FTC/TAF (Genvoya) or EVG/COBI/FTC/TDF (Stribild);
4. HIV is currently suppressed, defined as:

   1. Plasma HIV-1 RNA <50 c/mL for ≥3 months preceding Screening; AND
   2. Plasma HIV-1 RNA <50 copies/mL at the Screening assessment; INCL 5. Documentation that the participant is negative for the human leukocyte antigen (HLA)-B*5701 allele.

Exclusion Criteria:

1. Pregnant, breastfeeding, or planning to become pregnant during the study period;
2. Bilateral hip replacement;
3. Exceeds weight limit for DEXA equipment (i.e., weighs >350 lbs or >159 kg);
4. History or presence of allergy to the study treatment (Triumeq) or any of its components (to ABC, DTG, or 3TC);
5. Active Centers for Disease Control and Prevention (CDC) Category C HIV-1 disease (see Section 17.1 for definition), with the exception of cutaneous Kaposi's sarcoma, not requiring systemic therapy and historic CD4+ cell counts of <200 cells/mm3;
6. Positive for hepatitis B virus surface antigen (HBsAg) at Screening;
7. Ongoing malignancies (other than localized malignancies, such as cutaneous Kaposi's sarcoma, basal cell carcinoma, cervical intraepithelial neoplasia);
8. Significant suicidal risk in the investigator's opinion;
9. Metabolic disease;
10. Treatment with HIV immunotherapeutic vaccine within 90 days of Screening;
11. Radiation, cytotoxic chemotherapy, or any immunomodulator (that alters immune responses) within 28 days of Screening;
12. Exposure to any experimental drug or vaccine within 28 days or 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to first dose of study treatment on Day 1;
13. History of use of only mono or dual NRTI therapy prior to starting combination ART for the treatment of HIV infection (except that prior NRTI use for the purpose of pre-exposure prophylaxis [PrEP] or postexposure prophylaxis [PEP] is not excluded);
14. Became HIV-positive (i.e., had a detectable plasma HIV-1 viral load) while taking PrEP or PEP;
15. Documented resistance to any component of the study treatment (ABC, DTG, or 3TC) as indicated by either:

    1. Historical genotype in the participant's medical record; OR
    2. Genotype obtained by GenoSure Archive evaluation at Screening;
16. Any verified screening Grade 4 laboratory abnormality that in the investigator's opinion is clinically significant;
17. Moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification;
18. Either of the following liver chemistry elevations:

    1. Alanine amintotransferase (ALT) ≥5 x the upper limit of normal (ULN); OR
    2. ALT ≥3 x ULN and bilirubin ≥1.5 x ULN (with >35% direct bilirubin);
19. Creatinine clearance (CrCl) of <50 mL/min (calculated by CockroftGault equation)
20. QT interval corrected for heart rate according to Bazett's formula (QTcB) ≥450 msec or QTcB ≥480 msec for participants with bundle branch block;
21. Any other condition or substance use that in the opinion of the investigator places the participants at undue risk from participation in the study or that may negatively impact the integrity of the study analyses.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Percent change from Baseline at Week 48 in total hip BMD (measured by DEXA) | 48 Weeks
Percent change from Baseline at Week 48 in lumbar spine BMD (measured by DEXA) | 48 Weeks

OTHER OUTCOMES:
Change from Baseline in bone biomarkers for individuals switching to ABC/DTG/3TC | 96 Weeks
Change from baseline in bone mineral density (in lumbar spine and total hip) assessed by T-scores and Z-scores from Baseline in individuals switching to ABC/DTG/3TC | 96 Weeks
  Z-score = (Patient's BMD - expected BMD) / SD; T-score = (BMD-Reference BMD)/SD Units are numerical in value. BMD)/SD Units are numerical in value.
Number of adverse events (including long-term virologic/immunologic responses, abnormal laboratory values, or untoward medical conditions) for individuals switching to ABC/DTG/3TC | 96 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony M Mills, MD, Principal Investigator — Mills Clinical Research
Locations (1):
- Mills Clinical Research, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes